CLINICAL TRIAL: NCT00461825
Title: Efficacy and Safety of Maintenance Neoral Compared to Bitherapy Neoral-Imurel or Neoral-CellCept in Renal Transplantation
Brief Title: Maintenance Neoral Monotherapy Compared to Bitherapy in Renal Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Afssaps-980654
Record Dates: First submitted 2007-03-30; First posted 2007-04-18 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Kidney Transplantation
Keywords: Immunosuppression; Kidney transplantation; multicenter study
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cyclosporin A: C0: 75-125ng/ml-dose adapted in the 3 groups
Drug: Group A: CsA + Azathioprine(1 to 2 mg/kg/day)
Drug: Group B: CsA + CellCept(500 mg x 2/day)
Drug: Group C: CsAm

SUMMARY:
We have previously defined factors that predict the long term success of maintenance CsA monotherapy (CsAm) after kidney transplantation : donor age < 40 years, serum creatinine level at the initiation of CsAm £ 125 µmol/L, no rejection episode before CsAm initiation. We have also shown that the 8-year graft survival in 329 selected patients enrolled in maintenance CsA-m was 84 % (Hurault de Ligny et al, Transplantation, 2000 ; 69 : 1327-1332). These results were obtained with an old formulation of cyclosporin, azathioprine, steroid withdrawal over the first year and induction antibody. This prospective randomized multicentre study was designed to clarify whether maintenance Neoral + MMF or Neoral + AZA is better than a CsAm and wether Neoral + MMF is better than Neoral + AZA in low immunological risk cadaveric kidney transplant recipients.

DETAILED DESCRIPTION:
Between july 1998 and january 2004 selected patients were randomly assigned equally within each centre to receive CsAm or bitherapy with equally CsA + MMF or CsA + AZA.

ELIGIBILITY:
* Inclusion criteria:

  * Primary cadaveric renal transplant with induction therapy, delayed Neoral, MMF and prednisone
  * Steroid withdrawal >= 3 months before enrolment
  * Bitherapy Neoral + CellCept
  * Follow up time since transplantation : 11-24 months
  * Recipient age >= 25 years
  * Donor age <= 45 years
  * Serum creatinine level <= 125 µmol/L and/or calculated creatinine clearance >= 50 ml/mn (CG formula)
  * No or only one steroid-sensitive acute rejection episode during the first year post-transplantation
  * PRA <= 25 %
  * Written informed consent
* Exclusion Criteria:

  * Living donor transplantation
  * Recipient receiving tacrolimus
  * Azathioprine intolerance
  * Thrombopenia < 100 000/mm³
  * Neutropenia < 1500/mm³
  * Hemoglobinemia <= 8g/dl
  * On going infection

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207
Dates: Start 1998-07; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
to compare maintenance CsAm with dual therapy groups and within dual therapy MMF with AZA for :
The incidence and the delay of occurrence of graft dysfunction episode defined as ³ 20 % increase in serum creatinine level (mean of three results obtained in the same laboratory) and requiring a graft biopsy.
Causes of graft dysfunction episodes diagnosed by graft biopsy.
The incidence of serious infections (HVZ, EBV, HPV genital infection, febrile UTI, pneumonitis...)

SECONDARY OUTCOMES:
To compare the three treatment groups for the following parameters :
Incidence of therapeutic failure defined by biopsy proven acute rejection episode or CsA renal toxicity
Graft function evaluated by serum creatinine level and calculated creatinine clearance (CG formula)
Adverse events
Patient and graft survival

CONTACTS AND LOCATIONS:
Overall Officials: TOUCHARD Guy, MD,Professor, Principal Investigator — Poitiers University Hospital, POITIERS, 86021, FRANCE
Locations (5):
- France (5):
  - Caen university Hospital, Caen
  - Dupuytren University Hospital, Limoges
  - Poitiers University hospital, Poitiers
  - Reims University Hospital, Reims
  - Rouen University Hospital, Rouen

REFERENCES:
- [Background] Hurault de Ligny B, Toupance O, Lavaud S, Bauwens M, Peyronnet P, Le Meur Y, Ryckelynck JP, Jolly D, Leroux-Robert C, Touchard G. Factors predicting the long-term success of maintenance cyclosporine monotherapy after kidney transplantation. Transplantation. 2000 Apr 15;69(7):1327-32. doi: 10.1097/00007890-200004150-00019. PMID 10798748
- [Background] Touchard G, Hauet T, Cogny Van Weydevelt F, Hurault de Ligny B, Peyronnet P, Lebranchu Y, Toupance O, N'Doye P, Busson M. Maintenance cyclosporin monotherapy after renal transplantation--clinical predictors of long-term outcome. Nephrol Dial Transplant. 1997 Sep;12(9):1956-60. doi: 10.1093/ndt/12.9.1956. PMID 9306349